CLINICAL TRIAL: NCT00755391
Title: Cognitive Behavioral Therapy for Adolescents With Bulimia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4819
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Bulimia Nervosa
Keywords: BN and subthreshold BN
MeSH Terms: conditions — Bulimia Nervosa | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- supportive psychotherapy (Placebo Comparator): supportive psychotherapy: 14 sessions
  Interventions: Behavioral: Supportive Psychotherapy
- cognitive behavior therapy (Active Comparator): cognitive behavior therapy: 14 sessions
  Interventions: Behavioral: cognitive behavior therapy

INTERVENTIONS:
Behavioral: cognitive behavior therapy — The cognitive behavioral therapy used in this study will focus on developing patterns of regular eating, addressing body image issues, and ways to cope with situations that trigger eating disordered behaviors.
  Arms: cognitive behavior therapy
Behavioral: Supportive Psychotherapy — The supportive psychotherapy treatment used in this study will involve identifying issues underlying your child's eating disorder and giving your child information about the psychological processes that tend to maintain or continue eating disorder symptoms.
  Arms: supportive psychotherapy

SUMMARY:
This pilot study will evaluate the effectiveness of individual cognitive behavioral therapy (CBT) and supportive psychotherapy (SP) in reducing bulimic symptoms among adolescents.

DETAILED DESCRIPTION:
Patients will be randomized to have an equal chance of either receiving CBT or SP. Participants will include both individuals with DSM-IV bulimia nervosa (BN), and patients with sub-threshold BN. Adolescent patients will be treated at the New York State Psychiatric Institute, with a target recruitment of 20 patients completing the study. Participants in both conditions will be assessed prior to treatment and at the end of treatment. This trial is intended to serve as a pilot investigation to determine the feasibility and utility of a larger controlled study in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 12 and 18
2. DSM-IV diagnosis of bulimia nervosa or sub-threshold bulimia nervosa (binge eating and/or purging at least once per week)

Exclusion Criteria:

1. Diagnosis of bipolar disorder
2. Current psychosis
3. Drug or alcohol abuse in the past 3 months
4. Acute Suicidal Risk
5. Major depression producing significant functional impairment
6. Significant medical illness
7. Weight outside of normal weight range (between 85% and 120% of the 50th percentile for age as measured by standard growth charts)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2008-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Examination scores | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Sysko, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States